CLINICAL TRIAL: NCT02789033
Title: Efficacy of the Combination of Isosorbide Dinitrate Spray and Chitosan in Diabetic Foot Ulcers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Leonel Garcia Benavides, Professor researcher, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 030-2010
Record Dates: First submitted 2015-03-24; First posted 2016-06-02 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Diabetic Foot Ulcers
Keywords: diabetic foot ulcers; chitosan; isosorbide dinitrate spray
MeSH Terms: conditions — Diabetic Foot | interventions — Chitosan; Polymers; Isosorbide Dinitrate; Glutathione Transferase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Chitosan (Active Comparator): Chitosan chemically is a high-molecular-weight linear polycationic heteropolysaccharide comprising copolymers of 1,4-linked D-glucosamine and N-acetyl-D-glucosamine
  Interventions: Drug: Chitosan; Drug: Isosorbide dinitrate
- Isosorbide dinitrate spray (Active Comparator): Isosorbide dinitrate spray (2.5 mg) is an organic nitrate, is a vasodilator with effects on both arteries and veins. The chemical name of ISDN is 1,4:3,6-dianhydro-D-glucitol 2,5-dinitrate.
  Interventions: Drug: Chitosan; Drug: Isosorbide dinitrate
- Placebo (Placebo Comparator): Placebo in the same pharmacological presentation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chitosan — Chitosan chemically is a high-molecular-weight linear polycationic heteropolysaccharide comprising copolymers of 1,4-linked D-glucosamine and N-acetyl-D-glucosamine
  Other Names: polymers
  Arms: Chitosan; Isosorbide dinitrate spray
Drug: Isosorbide dinitrate — Isosorbide dinitrate (ISDN), is an organic nitrate, is a vasodilator with effects on both arteries and veins. The chemical name of ISDN is 1,4:3,6-dianhydro-D-glucitol 2,5-dinitrate
  Other Names: organic nitrate
  Arms: Chitosan; Isosorbide dinitrate spray
Drug: Placebo — placebo
  Other Names: Magnessium Calcuim
  Arms: Placebo

SUMMARY:
The prevalence of diabetic foot ulceration in the diabetic population is 4-10%; the condition is more frequent in elder patients. It is estimated that about 5% of all patients with diabetes present a history of foot ulceration, while the lifetime risk of diabetic patients developing this complication is 15%. The majority (60-80%) of foot ulcers will heal, while 10-15% of them will remain active, and 5-24% of them will finally lead to limb amputation within a period of 6-18 months after the first evaluation , 2 out of 3 patients with a limb amputation could also be involved in a new amputation in the next year; higher or in the other leg , Eighty-five percent of lower-limb amputations in patients with diabetes are preceded by foot ulceration. The management of chronic diabetic foot ulcers (DFU) suggests multi-disciplinary approaches including control of diabetes, orthotic shoe wear, off-loading device, wound care and surgery in selected cases. However, treatment of DFU remains challenging because of unsatisfactory results from surgical and non-surgical treatments. Many adjunctive therapies are designed to improve the care of DFU including negative pressure wound therapy , ultrasound, recombinant human platelet-derived growth factor-BB (rPDGF-BB) Hyperbaric oxygen and acellular matrix product among others.

DETAILED DESCRIPTION:
A randomized, placebo controlled, double-blind Clinical trial was designed. 60 Patients with diabetic foot ulcers in grade I and II of the classification of Wagner, with leg arm index> 0.8 and without specific treatment for foot ulcers referred to the experimental and clinical Therapeutic Institute will be included. All patients give written informed consent; previously the protocol was approved for the bioethics committee of the CUCS, of the Guadalajara University, registration number 030-2010. Patients with another type of topical medication will be excluded. Isosorbide dinitrate spray (2.5 mg).

Preparation of chitosan Hydrogels: The composition of gel formulation will be given prior training. ISDN and chitosan gel will be applied handled under aseptic conditions to the wound, and covered with sterile bandages. The patients will be evaluated every 2 weeks (macroscopic study and measurement of the ulcerated area) until 6 views. A second biopsy will be done one week before the finalization of the treatment of 15 weeks. The biopsies will be embedded on paraformaldehyde (4%) and paraffin. Sections of 5 µm were analyzed by a pathologist to determine hypertrophic and hyperplasic capillaries, inflammation and cellular matrix using Hematoxylin & eosin and Masson's trichrome stains. An immunohistochemical stain was also realized to evaluate several molecular markers such as α-SMA (abcam, Cambridge, MA), Desmin (abcam, Cambridge, MA), VEGF (abcam, Cambridge, MA) and Von Willebrand Factor (Chemicon, CA). (figure 1) Statistical analysis: It will be done using SPSS program for Windows Version 10.0, the results of quantitative variables were expressed in average and standard deviation. The differences between baseline and subsequent pharmacologic intervention measurements will be investigated with the Wilcoxon test. The Mann Whitney U test will be used to compare groups. Frequencies by categories as well as percentages will be quantified for qualitative variables. Comparisons between groups were performed with Chi2. For all comparisons p < 0.05 will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetic foot ulcers in grade I and II of the classification of Wagner
* with leg arm index> 0.8 and
* without specific treatment for foot ulcers referred to the experimental and clinical

Exclusion Criteria:

* Patients with another type of topical medication
* patients with diabetic foot ulcers in grade III and
* with leg arm index <0.8

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonel Garcia, PhD, Principal Investigator — University of Guadalajara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexiadou K, Doupis J. Management of diabetic foot ulcers. Diabetes Ther. 2012 Nov;3(1):4. doi: 10.1007/s13300-012-0004-9. Epub 2012 Apr 20. PMID 22529027
- [Background] Reiber GE, Lipsky BA, Gibbons GW. The burden of diabetic foot ulcers. Am J Surg. 1998 Aug;176(2A Suppl):5S-10S. doi: 10.1016/s0002-9610(98)00181-0. PMID 9777967
- [Background] Xie X, McGregor M, Dendukuri N. The clinical effectiveness of negative pressure wound therapy: a systematic review. J Wound Care. 2010 Nov;19(11):490-5. doi: 10.12968/jowc.2010.19.11.79697. PMID 21135797
- [Background] Tiaka EK, Papanas N, Manolakis AC, Maltezos E. The role of hyperbaric oxygen in the treatment of diabetic foot ulcers. Angiology. 2012 May;63(4):302-14. doi: 10.1177/0003319711416804. Epub 2011 Aug 25. PMID 21873346
- [Background] Schaffer MR, Tantry U, Efron PA, Ahrendt GM, Thornton FJ, Barbul A. Diabetes-impaired healing and reduced wound nitric oxide synthesis: a possible pathophysiologic correlation. Surgery. 1997 May;121(5):513-9. doi: 10.1016/s0039-6060(97)90105-7. PMID 9142149
- [Background] Andrews KL, Irvine JC, Tare M, Apostolopoulos J, Favaloro JL, Triggle CR, Kemp-Harper BK. A role for nitroxyl (HNO) as an endothelium-derived relaxing and hyperpolarizing factor in resistance arteries. Br J Pharmacol. 2009 Jun;157(4):540-50. doi: 10.1111/j.1476-5381.2009.00150.x. Epub 2009 Mar 26. PMID 19338582
- [Background] Raafat D, von Bargen K, Haas A, Sahl HG. Insights into the mode of action of chitosan as an antibacterial compound. Appl Environ Microbiol. 2008 Jun;74(12):3764-73. doi: 10.1128/AEM.00453-08. Epub 2008 May 2. PMID 18456858
- [Background] Sezer AD, Cevher E, Hatipoglu F, Ogurtan Z, Bas AL, Akbuga J. Preparation of fucoidan-chitosan hydrogel and its application as burn healing accelerator on rabbits. Biol Pharm Bull. 2008 Dec;31(12):2326-33. doi: 10.1248/bpb.31.2326. PMID 19043221
- [Background] Girach A, Manner D, Porta M. Diabetic microvascular complications: can patients at risk be identified? A review. Int J Clin Pract. 2006 Nov;60(11):1471-83. doi: 10.1111/j.1742-1241.2006.01175.x. PMID 17073842
- [Background] Chabbert-Buffet N, LeDevehat C, Khodabandhelou T, Allaire E, Gaitz JP, Tribout L, Abdoucheli-Baudot N, Vayssairat M. Evidence for associated cutaneous microangiopathy in diabetic patients with neuropathic foot ulceration. Diabetes Care. 2003 Mar;26(3):960-1. doi: 10.2337/diacare.26.3.960. No abstract available. PMID 12610079
- [Background] Richards AM, Floyd DC, Terenghi G, McGrouther DA. Cellular changes in denervated tissue during wound healing in a rat model. Br J Dermatol. 1999 Jun;140(6):1093-9. doi: 10.1046/j.1365-2133.1999.02908.x. PMID 10354076

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: ADDITIONAL PARTICIPANTS WERE INCLUDED ANTICIPATING PARTICIPANTS WHO DO NOT COMPLETE THE CLINICAL TRIAL
Groups:
- Active Comparator: Chitosan: Chitosan chemically is a high-molecular-weight linear polycationic heteropolysaccharide comprising copolymers of 1,4-linked D-glucosamine and N-acetyl-D-glucosamine
  And
  Placebo in the same pharmacological presentation that Isosorbide dinitrate spray
- Active Comparator: Isosorbide Dinitrate Spray: Isosorbide dinitrate spray (2.5 mg) is an organic nitrate, is a vasodilator with effects on both arteries and veins. The chemical name of ISDN is 1,4:3,6-dianhydro-D-glucitol 2,5-dinitrate.
  And
  Placebo in the same pharmacological presentation that Chitosan
- Combination: IDS and Chitosan: Isosorbide dinitrate spray (2.5 mg) is an organic nitrate, is a vasodilator with effects on both arteries and veins. The chemical name of ISDN is 1,4:3,6-dianhydro-D-glucitol 2,5-dinitrate.
  And
  Chitosan chemically is a high-molecular-weight linear polycationic heteropolysaccharide comprising copolymers of 1,4-linked D-glucosamine and N-acetyl-D-glucosamine
- Placebo Comparator: Placebo: Placebo in the same pharmacological presentation that both, IDS and Chitosan.
Period: Overall Study
Arm/Group | Active Comparator: Chitosan | Active Comparator: Isosorbide Dinitrate Spray | Combination: IDS and Chitosan | Placebo Comparator: Placebo
Started | 17 | 17 | 17 | 17
Completed | 15 | 15 | 16 | 15
Not Completed | 2 | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator: Chitosan | Active Comparator: Isosorbide Dinitrate Spray | Combination: IDS and Chitosan | Placebo Comparator: Placebo | Total
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 17 | 17 | 68
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 8 | 8 | 32
  Male | 9 | 9 | 9 | 9 | 36
Diameter of the ulcer [Mean (Standard Deviation); unit: centimeters] | 10.5 (5.8) | 12.1 (7.0) | 11.4 (8.2) | 15.8 (9.3) | 12.3 (7.5)

OUTCOME MEASURES:

1. Primary Outcome: Biopsies
Description: Histological changes in ulcers
Time Frame: 75 days
Measure: Mean (Standard Deviation); unit: UI/dL
Arm/Group | Active Comparator: Chitosan | Active Comparator: Isosorbide Dinitrate Spray | Combination: IDS and Chitosan | Placebo Comparator: Placebo
Number analyzed (Participants) | 15 | 15 | 16 | 15
UI/dL
  α-smooth muscle actin | 2.46 (0.6) | 2.64 (0.6) | 2.56 (0.6) | 2.07 (0.6)
  Von Willebrand Factor | 2.38 (0.65) | 2.28 (0.82) | 2.31 (0.8) | 2.15 (0.5)
  vascular endothelial growth factor-A | 2.23 (0.8) | 2.6 (0.6) | 2.43 (0.6) | 2.07 (0.7)
  desmin | 2.3 (0.8) | 2.5 (0.6) | 2.6 (0.6) | 2.3 (0.6)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Chitosan and isosorbide dinitrate are widely used substances, in addition they were used in regular doses for a short period of time, locally.
Arm/Group | Active Comparator: Chitosan | Active Comparator: Isosorbide Dinitrate Spray | Combination: IDS and Chitosan | Placebo Comparator: Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No